CLINICAL TRIAL: NCT00048841
Title: Prevention of Osteoporosis in Men With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: DK61535 (completed)
Record Dates: First submitted 2002-11-08; First posted 2002-11-13 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Prostate Cancer; Osteoporosis; Hypogonadism
Keywords: Male; Osteoporosis; Prostate cancer; Hypogonadism; Bisphosphonates; Bone mineral density
MeSH Terms: conditions — Prostatic Neoplasms; Osteoporosis; Hypogonadism | interventions — Alendronate

INTERVENTIONS:
Drug: alendronate

SUMMARY:
The purpose of this two year study is to examine the safety and effectiveness of alendronate (Fosamax) for the prevention of bone loss in men with prostate cancer who are on therapy to lower their testosterone levels. All men will receive appropriate calcium and vitamin D supplements and one to two years of alendronate therapy. Bone density tests will be done every six months.

DETAILED DESCRIPTION:
Prostate cancer is the most common visceral malignancy and second leading cause of cancer death in men. While androgen ablation therapy is the cornerstone of treatment for more advanced stage disease, recent studies suggest the advantage of introducing androgen deprivation much earlier. Because androgens are essential in maintaining skeletal integrity in men, androgen deprivation therapy constitutes a major risk factor for male osteoporosis. We have previously demonstrated that men on chronic androgen deprivation therapy have up to 20% loss of bone. Our hypotheses are that: 1) chronically increased bone resorption induced by long term androgen deprivation therapy in men with prostate cancer can be reversed with once weekly bisphosphonate; 2) the improvement in bone mass with bisphosphonate therapy will be reflected by changes in biochemical markers of bone turnover and will allow us to predict who will respond to therapy; and 3) following termination of bisphosphonate therapy, bone mass will be maintained despite the absence of antiresorptive therapy. To address these hypotheses, we will enroll 84 men with stage D0 prostate cancer who have been on chronic androgen deprivation therapy in a two year, double blind, placebo controlled, randomized, modified crossover clinical design. During the first year, subjects will be randomized to bisphosphonate therapy or placebo. During the second year, all subjects who were on placebo will receive active treatment and all subjects who were on active treatment will be randomly assigned to continue therapy or change to placebo. To evaluate the effect of bisphosphonate on preventing bone loss, we will assess bone mass of the spine, total hip, total body, and forearm by dual-energy X-ray absorptiometry. For hypothesis 2, we will assess markers of bone resorption and formation to determine if early changes in markers are associated with long term changes in bone mass. For hypothesis 3, we will continue to follow bone mass and biochemical markers of bone turnover between months 12 and 24 to examine rates of change when antiresorptive therapy is terminated. Few data are available on the prevention of bone loss in men on androgen deprivation therapy. This study will examine a preventive strategy, the potential mechanism of bone loss, the ability of biochemical markers to predict bone mass, and skeletal outcomes when antiresorptive therapy is withdrawn.

ELIGIBILITY:
Inclusion Criteria:

* Men age 50-85
* Stage D0 prostate cancer
* On androgen deprivation therapy

Exclusion Criteria:

* Renal failure
* Hyperthyroidism
* Cushing's syndrome
* Metabolic bone disease
* Use of glucocorticoids
* Use of certain anticonvulsants
* On osteoporosis therapies
* Nonprostate cancers

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112
Dates: Start 2002-05; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
PA spine BMD over 1 year
Change in PA spine BMD over 2nd year

SECONDARY OUTCOMES:
BMD at the hip and lateral spine

CONTACTS AND LOCATIONS:
Overall Officials: Susan L. Greenspan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Osteoporosis Prevention & Treatment Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Greenspan SL, Nelson JB, Trump DL, Resnick NM. Effect of once-weekly oral alendronate on bone loss in men receiving androgen deprivation therapy for prostate cancer: a randomized trial. Ann Intern Med. 2007 Mar 20;146(6):416-24. doi: 10.7326/0003-4819-146-6-200703200-00006. PMID 17371886